CLINICAL TRIAL: NCT03912337
Title: Effect of Erenumab-aooe on Disability and Work Productivity in Employed Subjects With Episodic Migraine Who Have Previously Failed 1 or More Migraine Preventive Treatments.
Brief Title: Effect of Erenumab-aooe on Disability and Work Productivity in Employed Subjects With Episodic Migraine
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated [Study would not complete enrollment target until 2026 with results available in 2027. The information will not be useful at that time.]
Sponsor: Amgen (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20180060
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Results first posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Migraine
Keywords: Episodic migraine; Disability; Migraine-related disability; Work productivity; Erenumab; AIMOVIG
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): After subjects complete baseline and are found eligible, they will be enrolled and randomized in a 1:1 ratio to either erenumab or placebo.
  Interventions: Drug: Placebo
- Erenumab (Experimental): After subjects complete baseline and are found eligible, they will be enrolled and randomized in a 1:1 ratio to either erenumab or placebo.
  Interventions: Drug: Erenumab

INTERVENTIONS:
Drug: Placebo — Placebo once every 4 weeks. SC injection.
  Arms: Placebo
Drug: Erenumab — Erenumab once every 4 weeks. SC injection.
  Other Names: Aimovig
  Arms: Erenumab

SUMMARY:
To evaluate the effect of erenumab compared to placebo on disability in employed subjects with episodic migraine (EM) who have previously failed 1 or more migraine preventive treatments.

DETAILED DESCRIPTION:
Migraine prevention continues to be an area of large, unmet medical need, with existing therapies often having modest efficacy and poor tolerability. Calcitonin gene-related peptide (CGRP) has an important role in the pathophysiology of migraine. Erenumab-aooe is a fully human monoclonal antibody that targets the CGRP receptor, and interrupts its downstream effects. Erenumab has been approved for the preventive treatment of migraine in adults. The present study is a Phase IV trial that will assess the effect of erenumab on disability and work productivity in employed subjects with episodic migraine (EM) who have previously failed 1 or more migraine preventive treatments.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age upon entry into screening.
* Documented history of migraine with or without aura according to the IHS ICHD-III for greater than or equal to 12 months
* Has EM defined as history of greater than or equal to 4 and less than 15 migraine days and less than 15 headache days per month on average during the 3 months prior to initial screening
* Employed greater than or equal to 20 hours/week upon entry into initial screening, stable for at least 3 months in the same job and has not specified willful termination of employment throughout the duration of the study. Employment is defined by work outside the home, self-employed, or works from home
* Has greater than or equal to 4 hours of lost productive time due to headache/migraine and/or related symptoms in the past month prior to initial screening as determined by subject
* Has total disability score of greater than 10 as assessed by MIDAS (3-month recall) at initial screening
* History of treatment failure with at least 1 preventive treatment category for migraine

Exclusion Criteria:

* Older than 50 years of age at migraine onset
* History of cluster headache, hemiplegic migraine, or other trigeminal autonomic cephalalgia.
* Taken an opioid and/or opioid-containing analgesic greater than or equal to 4 days during the 1 month prior to screening for any indication
* Taken a butalbital and/or butalbital-containing analgesic greater than or equal to 4 days during the 1 month prior to screening for any indication
* Change in the regimen of current migraine preventive treatment or a concomitant medication that may have migraine prevention effects during baseline
* Taken an opioid and/or opioid-containing analgesic ≥ 4 days during baseline for any indication.
* Taken a butalbital and/or butalbital-containing analgesic ≥ 4 days during baseline for any indication.
* Previously treated with any agent (monoclonal antibody or small molecule) targeting the CGRP pathway (ligand or receptor) in preventive settings

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (28):
- United States (28):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Los Angeles, California
  - Research Site, Pasadena, California
  - Research Site, Basalt, Colorado
  - Research Site, East Hartford, Connecticut
  - Research Site, New London, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Jacksonville, Florida
  - Research Site, Orlando, Florida
  - Research Site, Chalmette, Louisiana
  - Research Site, Hagerstown, Maryland
  - Research Site, Worcester, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Bolivar, Missouri
  - Research Site, City of Saint Peters, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Toms River, New Jersey
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Centerville, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Frisco, Texas
  - Research Site, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 13 centers in the United States of America. The study consisted of a 4-week baseline period and a 6-month double-blind treatment period (DBTP).
Pre-assignment Details: Eligible participants were randomized in a 1:1 ratio to either erenumab 140 milligrams (mg) or placebo once monthly (QM).
Groups:
- Placebo QM: Participants randomized to receive placebo QM for 6 months during the DBTP.
- Erenumab 140 mg QM: Participants randomized to receive erenumab 140 mg QM for 6 months during the DBTP.
Period: Overall Study
Arm/Group | Placebo QM | Erenumab 140 mg QM
Started | 15 | 14
Completed | 13 | 13
Not Completed | 2 | 1
Not completed — Withdrawal of Consent From Study | 1 | 0
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: The respective full analysis set consisted of all participants who were randomized in the study through traditional study sites or decentralized clinical trial sites (DCTS).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QM | Erenumab 140 mg QM | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (9.9) | 38.6 (15.4) | 39.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 13 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 14 | 27
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Modified Migraine Disability Assessment (MIDAS) Total Score [Mean (Standard Deviation); unit: score on a scale] — The modified MIDAS Questionnaire is a 5-item questionnaire that measures headache-related disability as lost time from paid work or school, housework, and non-work (family, social, and leisure) activities. Participants provided the number of productive days lost or productivity reduced by half or more over the past month due to headache (item score range from 0 to 31). Productive days lost counted in items 1 and 3 were not included for items 2 and 4, respectively. The 5 item scores were summed to calculate the MIDAS total score (range from 0 to 93). Higher scores indicated a worse outcome.
  score on a scale | 20.3 (11.5) | 23.1 (11.3) | 21.7 (11.3)
Monthly Migraine Days (MMD) [Mean (Standard Deviation); unit: migraine days per month] — A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache) or received migraine-specific medication during aura. A qualified migraine headache was defined either as a migraine (≥30 minutes) with or without aura.
  MMD were calculated as the number of migraine days in the 4-week baseline period.
  migraine days per month | 9.2 (3.7) | 9.0 (2.8) | 9.1 (3.2)
Monthly Percent Work Impairment [Mean (Standard Deviation); unit: percentage of monthly workdays impaired] — Percent work impairment was calculated based on questions 2, 4 and 5 of the Work Productivity and Activity Impairment (WPAI) Migraine-Questionnaire and could range from 0% to 100%. The questionnaire was collected weekly. The monthly percent work impairment was equal to the arithmetic mean of the observed weekly percent work impairment over the monthly interval (4-week baseline period). Higher scores indicate greater impairment.
  percentage of monthly workdays impaired | 49.5 (19.0) | 57.6 (13.5) | 53.4 (16.8)
Migraine Functional Impact Questionnaire (MFIQ) - Impact on Physical Functioning Domain Score [Mean (Standard Deviation); unit: score on a scale] — The MFIQ is a self-administered 26-item instrument measuring the impact of migraine on broader functioning. Participants responded to 5 items in the impact on physical functioning domain using a 5-point scale assigned scores from 1 to 5, with 5 representing the greatest burden. The scores were calculated as the sum of the item responses rescaled to a 0 to 100 scale, with higher scores representing greater impact of migraine, i.e., higher burden.
  score on a scale | 46.5 (17.9) | 56.8 (23.8) | 51.5 (21.2)
MFIQ - Impact on Usual Activities Domain Score [Mean (Standard Deviation); unit: score on a scale] — The MFIQ is a self-administered 26-item instrument measuring the impact of migraine on broader functioning. Participants responded to 10 items in the impact on usual activities domain using a 5-point scale assigned scores from 1 to 5, with 5 representing the greatest burden. The scores were calculated as the sum of the item responses rescaled to a 0 to 100 scale, with higher scores representing greater impact of migraine, i.e., higher burden.
  score on a scale | 38.5 (15.5) | 51.3 (20.0) | 44.7 (18.6)
MFIQ - Impact on Social Functioning Domain Score [Mean (Standard Deviation); unit: score on a scale] — The MFIQ is a self-administered 26-item instrument measuring the impact of migraine on broader functioning. Participants responded to 5 items in the impact on social functioning domain using a 5-point scale assigned scores from 1 to 5, with 5 representing the greatest burden. The scores were calculated as the sum of the item responses rescaled to a 0 to 100 scale, with higher scores representing greater impact of migraine, i.e., higher burden.
  score on a scale | 41.8 (18.6) | 54.2 (19.4) | 47.8 (19.7)

OUTCOME MEASURES:

1. Primary Outcome: Sum of Monthly Changes From Baseline in Modified MIDAS Total Score Over the 6-month DBTP
Description: The modified MIDAS Questionnaire is a 5-item questionnaire that measures headache-related disability as lost time from paid work or school, housework, and non-work (family, social, and leisure) activities. Participants provided the number of productive days lost or productivity reduced by half or more over the past month due to headache (item score range from 0 to 31). Productive days lost counted in items 1 and 3 were not included for items 2 and 4, respectively. The 5 item scores were summed to calculate the MIDAS total score (range from 0 to 93). The change from baseline was calculated by subtracting the baseline total score from the total score calculated each month. The change from baseline values for Months 1 to 6 were then summed to calculate the sum of monthly changes from baseline (range from -558 to 558). A negative sum of changes from baseline indicated a better outcome.
Time Frame: Baseline and Months 1 to 6
Population: The respective efficacy analysis set (EAS) consisted of a subset of participants from traditional study sites or DCTS who received at least 1 dose of investigational product (IP) and had a baseline value and at least 1 post baseline value for the endpoint of interest. Participants were analyzed according to their randomized treatment, regardless of the treatment received.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo QM | Erenumab 140 mg QM
Number analyzed (Participants) | 15 | 14
score on a scale | -71.17 (60.81) | -98.03 (71.04)

2. Secondary Outcome: Change From Baseline in Mean MMD Over Months 4, 5, and 6 of the 6-month DBTP
Description: A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache) or received migraine-specific medication during aura. A qualified migraine headache was defined either as a migraine (≥30 minutes) with or without aura.
  The change from baseline in monthly migraine days was calculated as the average number of migraine days per month during the last 3 months (months 4, 5, and 6) of the 24-week double-blind treatment phase subtract the number of migraine days during the 4-week baseline phase. A negative change from baseline indicates a better outcome.
Time Frame: Baseline and the last 3 months (months 4, 5, and 6) of the 6-month DBTP
Population: The respective EAS including only participants with observed MMD data.
Measure: Mean (Standard Deviation); unit: migraine days per month
Arm/Group | Placebo QM | Erenumab 140 mg QM
Number analyzed (Participants) | 14 | 14
migraine days per month | -3.01 (2.51) | -5.60 (3.68)

3. Secondary Outcome: Change From Baseline in Mean Monthly Percent Work Impairment Over Months 4, 5, and 6 of the 6-month DBTP
Description: Percent work impairment was calculated based on questions 2, 4 and 5 of the Work Productivity and Activity Impairment (WPAI) Migraine-Questionnaire and could range from 0% to 100%. The questionnaire was collected weekly. The monthly percent work impairment was equal to the arithmetic mean of the observed weekly percent work impairment over the monthly interval. Higher scores indicate greater impairment.
  Change from baseline in mean monthly percent work impairment was calculated as the average of monthly percent work impairment over the last 3 months (month 4, 5, and 6) of the 24-week double-blind treatment phase minus the baseline score. A negative change from baseline indicates a better outcome.
Time Frame: Baseline and the last 3 months (months 4, 5, and 6) of the 6-month DBTP
Population: The respective EAS including only participants with observed WPAI data.
Measure: Mean (Standard Deviation); unit: percentage of monthly workdays impaired
Arm/Group | Placebo QM | Erenumab 140 mg QM
Number analyzed (Participants) | 14 | 12
percentage of monthly workdays impaired | -28.84 (14.55) | -31.72 (16.00)

4. Secondary Outcome: Change From Baseline in Mean MFIQ Physical Functioning Domain Score Over Months 4, 5, and 6 of the 6-month DBTP
Description: The MFIQ is a self-administered 26-item instrument measuring the impact of migraine on broader functioning. Participants responded to 5 items on the impact on physical functioning domain using a 5-point scale assigned scores from 1 to 5, with 5 representing the greatest burden. The scores were calculated as the sum of the item responses rescaled to a 0 to 100 scale, with higher scores representing greater impact of migraine, i.e., higher burden.
  The MFIQ physical functioning domain score was calculated per month for months 4, 5, and 6 and the mean over this period was calculated. The MFIQ physical functioning domain score during the 4-week baseline period was then subtracted to calculate the change from baseline in mean MFIQ physical functioning domain score over months 4, 5,and 6 of the 6-month DBTP. A negative change from baseline indicates a better outcome.
Time Frame: Baseline and the last 3 months (months 4, 5, and 6) of the 6-month DBTP
Population: The respective EAS including only participants with observed MFIQ data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo QM | Erenumab 140 mg QM
Number analyzed (Participants) | 14 | 13
score on a scale | -22.44 (18.62) | -31.99 (33.05)

5. Secondary Outcome: Change From Baseline in Mean MFIQ Usual Activities Domain Score Over Months 4, 5, and 6 of the 6-month DBTP
Description: The MFIQ is a self-administered 26-item instrument measuring the impact of migraine on broader functioning. Participants responded to 10 items on the impact on usual activities domain using a 5-point scale assigned scores from 1 to 5, with 5 representing the greatest burden. The scores were calculated as the sum of the item responses rescaled to a 0 to 100 scale, with higher scores representing greater impact of migraine, i.e., higher burden.
  The MFIQ usual activities domain score was calculated per month for months 4, 5, and 6 and the mean over this period was calculated. The MFIQ usual activities domain score during the 4-week baseline period was then subtracted to calculate the change from baseline in mean MFIQ usual activities domain score over months 4, 5,and 6 of the 6-month DBTP. A negative change from baseline indicates a better outcome.
Time Frame: Baseline and the last 3 months (months 4, 5, and 6) of the 6-month DBTP
Population: The respective EAS including only participants with observed MFIQ data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo QM | Erenumab 140 mg QM
Number analyzed (Participants) | 14 | 13
score on a scale | -20.82 (13.15) | -30.77 (25.50)

6. Secondary Outcome: Change From Baseline in Mean MFIQ Social Functioning Domain Score Over Months 4, 5, and 6 of the 6-month DBTP
Description: The MFIQ is a self-administered 26-item instrument measuring the impact of migraine on broader functioning. Participants responded to 5 items on the impact on social functioning domain using a 5-point scale assigned scores from 1 to 5, with 5 representing the greatest burden. The scores were calculated as the sum of the item responses rescaled to a 0 to 100 scale, with higher scores representing greater impact of migraine, i.e., higher burden.
  The MFIQ social functioning domain score was calculated per month for months 4, 5, and 6 and the mean over this period was calculated. The MFIQ social functioning domain score during the 4-week baseline period was then subtracted to calculate the change from baseline in mean MFIQ social functioning domain score over months 4, 5,and 6 of the 6-month DBTP. A negative change from baseline indicates a better outcome.
Time Frame: Baseline and the last 3 months (months 4, 5, and 6) of the 6-month DBTP
Population: The respective EAS including only participants with observed MFIQ data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo QM | Erenumab 140 mg QM
Number analyzed (Participants) | 14 | 13
score on a scale | -30.51 (21.15) | -41.44 (28.37)

ADVERSE EVENTS:
Time Frame: Baseline up to Month 6
Description: The respective safety analysis set consisted of all randomized participants from traditional study sites or DCTS who received at least 1 dose of IP.
Arm/Group | Placebo QM | Erenumab 140 mg QM
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 7/15 | 9/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QM (N=15) | Erenumab 140 mg QM (N=14)
Bradycardia (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Cyst (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
Infected dermal cyst (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dizziness postural (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 | 0
Generalised anxiety disorder (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0
Polymenorrhoea (Reproductive system and breast disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to slow enrollment and the impact of COVID-19 on the work productivity study endpoints, beyond normal operational disruptions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT03912337/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT03912337/SAP_001.pdf